CLINICAL TRIAL: NCT02301260
Title: Speed of Processing Training to Improve Cognition in Multiple Sclerosis: A Randomized Clinical Trial
Brief Title: Speed of Processing Training to Improve Cognition in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Neuropsychology and Neuroscience Laboratory, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RG 4997A5/1
Record Dates: First submitted 2014-04-23; First posted 2014-11-25 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis
Keywords: Processing Speed; Intervention; Multiple Sclerosis; Cognition
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Speed of Processing Training (SPT) (Experimental): SPT will be administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Interventions: Behavioral: Speed of Processing Training (SPT)
- Placebo control group (Placebo Comparator): Placebo control exercises will be administered on a laptop computer twice a week for 5 weeks (10 sessions)
  Interventions: Behavioral: Placebo Control

INTERVENTIONS:
Behavioral: Speed of Processing Training (SPT)
  Arms: Speed of Processing Training (SPT)
Behavioral: Placebo Control — Placebo control exercises will be administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Arms: Placebo control group

SUMMARY:
The purpose of this research study is to investigate the effectiveness of a computerized technique designed to improve processing speed (i.e. the amount of time it takes for a person's brain to process information) in a multiple sclerosis (MS) population. The study is designed to study how well this technique can help people with MS increase their processing speed and their ability to function better in everyday life. This treatment protocol has been studied extensively with older adults, showing improvements on standard laboratory measures of processing speed and performance of activities of daily living.

DETAILED DESCRIPTION:
This study is a double-blind, placebo-control randomized clinical trial examining the efficacy of Speed of Processing Training (SPT) for improving processing speed (PS) deficits in persons with Multiple Sclerosis (MS). Slowed PS is one of the most common deficits in individuals with MS and such deficits have been shown to exert significant negative impact on multiple aspects of everyday life, including occupational and social functioning. Despite these findings, few studies have attempted to remediate PS deficits in order to improve the everyday functioning of individuals with MS. This study is designed to (1) apply a treatment protocol for PS impairments well-validated in an aging population to individuals with MS with objectively observable deficits in PS and document its efficacy on standard neuropsychological outcome measures. In addition, the investigators will (2) assess the effectiveness of the intervention utilizing global measures of everyday life, including an objective measure (the Timed Activities of Daily Living; TIADL), as well as additional questionnaires to be completed by both the participant and a significant other. This study is also designed to (3) examine the influence of degree of PS impairment on treatment efficacy using neuropsychological tests, (4) evaluate the long-term effects of the treatment protocol and (5) examine the utility of booster sessions to facilitate long-term treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* English as a primary language
* diagnosis of Multiple Sclerosis
* processing speed impairment (based on evaluation)

Exclusion Criteria:

* most recent exacerbation within one month
* currently taking steroids or benzodiazepines
* history of significant psychiatric illness (bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder
* significant alcohol or drug abuse history

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change in scores on standardized tests of processing speed | Three points in time: baseline (week1), immediately following treatment (week 7) and 6 months after treatment is completed

SECONDARY OUTCOMES:
Change in scores on self-report of emotional functioning, measured via questionnaire | Three points in time: baseline (week1), immediately following treatment (week 7) and 6 months after treatment is completed
  Self-report questionnaires and objective measures of everyday performance will be used to determine whether there have been changes across the three time points.
Change in scores on self-report of everyday functioning, measured via questionnaire | Three points in time: pre-treatment, immediately following treatment and 6 months after treatment is completed
Change in scores on self-report of quality of life, measured via questionnaire | Three points in time: baseline (week1), immediately following treatment (week 7) and 6 months after treatment is completed

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chiaravalloti, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

REFERENCES:
- [Derived] Goverover Y, Costa S, DeLuca J, Chiaravalloti N. The Efficacy of the Speed of Processing Training Program in Improving Functional Outcome: From Restoration to Generalization. Arch Phys Med Rehabil. 2023 Jun;104(6):925-931. doi: 10.1016/j.apmr.2023.01.017. Epub 2023 Feb 8. PMID 36758712